#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for a single-centre, double-blind (sponsor open), placebo controlled two part study to evaluate the safety, tolerability and pharmacokinetics of single and repeat doses of GSK2292767 as a dry powder in healthy participants who smoke cigarettes. |
|---|---|---|
| <b>Compound Number</b> | : | GSK2292767 |
| Effective Date | : | 23-May-2017 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 202062.
- This RAP is intended to describe the safety, pharmacokinetic and exploratory pharmacodynamic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Statistician (Clinical Statistics) | NA | (Author) |
| Clinical Pharmacology | 19-May-2017 | Approval via E-mail |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Programming Manager (Respiratory Clinical Programming) | 15-May-2017 | E-mail |
| Data Quality Lead (Respiratory CPSSO Data Management) | 19-May-2017 | E-mail |
| Programmer/Analyst (Respiratory Clinical Programming) | 18-May-2017 | E-mail |
| Clinical Development Manager (Respiratory R&D Projects Clinical Platforms and Sciences) | 15-May-2017 | E-mail |
| Director of Human Translational Models and<br>Biomarkers (Respiratory TAU & Flexible<br>Discovery Unit) | 17-May-2017 | E-mail |
| Medical Director, SERM (Global Medical) | 16-May-2017 | E-mail |
| Head (Respiratory TAU & Flexible Discovery Unit) | 18-May-2017 | E-mail |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | <b>Approval Method</b> |
|------------------------------------|-------------|------------------------|
| Director, Statistics & Programming | 23-May-2017 | E-mail |
| Manager, Programming | 22-May-2017 | E-mail |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 6 |
| 2. | SUMN | ARY OF | KEY PROTOCOL INFORMATION | 7 |
| ۷. | 2.1. | | s to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | | bjective(s) and Endpoint(s) | |
| | ۷.۷. | Study O | bjective(s) and Endpoint(s) | |
| 3. | PI AN | NED ANA | ALYSES | 8 |
| Ο. | 3.1. | | Analyses | |
| | 3.2. | | alyses | |
| | 0.2. | i iiidi / tii | ury 000 | |
| 4. | ANAL' | YSIS POF | PULATIONS | 9 |
| | 4.1. | | Deviations | |
| 5. | HAND | LING CO | NVENTIONS | 10 |
| 6. | STUD | Y POPUL | ATION ANALYSES | 10 |
| | 6.1. | Overvie | w of Planned Analyses | 10 |
| 7. | | | TISTICAL ANALYSES | |
| | 7.1. | Safety A | Analyses | |
| | | 7.1.1. | Overview of Planned Safety Analyses | 11 |
| | | 7.1.2. | During the Study | 11 |
| | | | 7.1.2.1. Dose Escalations | |
| | | 7.1.3. | Final Safety Data | 12 |
| 8. | | | STATISTICAL ANALYSES | |
| | 8.1. | | cokinetic Analyses | |
| | | 8.1.1. | J | |
| | | 8.1.2. | Drug Concentration Measures | 13 |
| | | | 8.1.2.1. Overview of Planned Pharmacokinetic | |
| | | | Analyses for Drug Concentrations | |
| | | 8.1.3. | Pharmacokinetic Parameters | |
| | | | 8.1.3.1. Deriving Pharmacokinetic Parameters | |
| | | 8.1.4. | BAL Parameters | 14 |
| | | 8.1.5. | Single Dose Escalation (Part A) | |
| | | 0.4.0 | 8.1.5.1. Statistical Analysis of Dose Proportionality | |
| | | 8.1.6. | Repeat Dose (Part B) | 16 |
| | | | 8.1.6.1. Statistical Analysis of Dose Accumulation and | 47 |
| | | | Steady State | 17 |
| | | 0.4.7 | 8.1.6.2. Statistical Analysis of Peak to Trough Ratio | |
| | | 8.1.7. | Population Pharmacokinetic Analyses | |
| | 8.2. | | codynamic Analyses (Parts A and B) | |
| | | 8.2.1. | Overview of Planned Pharmacodynamic Analyses | |
| | | 8.2.2. | Planned Pharmacodynamic Statistical Analyses | 19 |
| 9. | REFE | RENCES | | 21 |
| 10. | | | | |
| | 10.1. | Appendi | ix 1: Time & Events | 23 |

#### CONFIDENTIAL

| 202062 |
|--------|
| 202062 |

| | 10.1.1. | Protocol De | efined Time & Events | 23 |
|---|---|---|---|---|
| | | | SOA – Part A (Single Dose) | |
| | | 10.1.1.2. | SOA – Part B (Repeat Dose) | 25 |
| 10.2. | Appendix | | ment Windows | |
| | 10.2.1. | <b>Definitions</b> | of Assessment Windows for Analyses | 28 |
| 10.3. | | | ent States and Phases | |
| | | | Phases | |
| | 10.3.2. | Treatment | States | 29 |
| | | | Treatment States for Concomitant Medication Data | 29 |
| | | | Treatment States for AE Data | |
| 10.4. | Appendix | | splay Standards & Handling Conventions | |
| | 10.4.1. | | tment & Sub-group Display Descriptors | |
| | 10.4.2. | | efinition & Derivations | |
| | | | Baseline Definitions | |
| | | | Derivations and Handling of Missing Baseline | |
| | | | Data | 31 |
| | 10.4.3. | | Process & Standards | |
| 10.5. | Appendix | | and Transformed Data | |
| | 10.5.1. | | | |
| | 10.5.2. | Study Popu | ulation | 33 |
| | 10.5.3. | Safety | | 34 |
| | 10.5.4. | Calculation | of Spirometry Screening Parameters | 35 |
| | 10.5.5. | Pharmacoo | dynamic | 35 |
| | 10.5.6. | Derivation | of BAL/ELF Drug Concentration Data | 36 |
| | 10.5.7. | Derivation | of BAL Cell Pellet Drug Concentration Data | 37 |
| 10.6. | Appendix | ι 6: Prematι | ure Withdrawals & Handling of Missing Data | 38 |
| | 10.6.1. | Premature | Withdrawals | 38 |
| | 10.6.2. | Handling of | f Missing Data | 38 |
| | | | Handling of Missing Dates | 39 |
| | | | Handling of Missing Data for Statistical | |
| | | | Analysis | |
| 10.7. | | | of Potential Clinical Importance | |
| | | • | Values | |
| | 10.7.2. | | | |
| | | | | 41 |
| 10.8. | Appendix | c 8: Model C | Checking and Diagnostics for Statistical | |
| | | | | 42 |
| | 10.8.1. | | Analysis Assumptions | |
| 10.9. | | | ion Pharmacokinetic Analyses | |
| | 10.9.1. | | ataset creation | |
| 10.10. | | | eviations & Trade Marks | |
| | | | ons | |
| | | | S | |
| 10.11. | | | Data Displays | |
| | | | ay Numbering | |
| | | | <del> –</del> | |
| | | | ulation Tables | |
| | | • | les | |
| | | | ıres | |
| | | | kinetic Tables | |
| | 10.11.7. | Pharmacok | kinetic Figures | 59 |

#### CONFIDENTIAL

| 10.11.8. Pharmacodynamic Tables | 6 <mark>2</mark> |
|---|---|
| 10.11.9. Pharmacodynamic Figures | 64 |
| 10.11.10. Pharmacokinetic / Pharmacodynamic Figures | |
| 10.11.11.ICH Listings: Part A (Single Dose Escalation) | |
| 10.11.12.ICH Listings: Part B (Repeat Dose) | <mark>70</mark> |
| 10.11.13. Non-ICH Listings: Part A (Single Dose Escalation) | 73 |
| 10.11.14. Non-ICH Listings: Part B (Repeat Dose) | 75 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe: Planned analyses and output for the final data. |
| Protocol | This RAP is based on Protocol Amendment 1(Dated: 05/JAN/2017) of study 202062 (GlaxoSmithKline Document Number 2016N288743_01) |
| Primary<br>Objective | To assess the safety and tolerability of single and repeat doses of GSK2292767 as a dry powder in healthy cigarette smokers. |
| Primary<br>Endpoint | Safety and tolerability of GSK2292767 as assessed by clinical monitoring of: Vital Signs Spirometry Electrocardiogram (ECG) Laboratory safety data Adverse events (AEs) |
| Study<br>Design | This is a two part, single site, randomised, double-blind (sponsor open), placebo controlled study in healthy smokers. |
| | Part A will consist of two 3-period interlocking cohorts. |
| | Part B is planned to follow Part A and is a parallel group design. The highest well tolerated dose achieved in Part A will be selected for Part B. |
| Planned<br>Analyses | All decisions regarding final analysis, as defined in this RAP document, will be made prior to Database Freeze (unblinding) of the study data. |
| Primary<br>Analysis<br>Population | Primary: Safety Population (Comprised of subjects who receive at least one dose of study treatment and will be based on the treatment which the subject actually received). |
| Estimation | An estimation and inference approach will be adopted to evaluate the objectives. |
| Primary<br>Analyses | Safety data will be presented in tabular and/or graphical format and summarised descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. |
| Secondary<br>Analyses | <ul> <li>Pharmacokinetic: Individual GSK2292767 plasma concentration-time profiles (by treatment and subject) and median/mean (±SD) profiles by treatment group will be plotted. Plasma concentration time data for GSK2292767 will be analyzed by non-compartmental methods using WinNonlin and derived PK parameters will be graphically presented, summarised and listed. Data will be analysed for dose proportionality and dose accumulation, peak to trough ratio and steady state.</li> <li>Pharmacodynamic: All endpoints will be presented in graphical format and/or</li> </ul> |
| | summarised descriptively and listed. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

One of the protocol defined endpoints was:

Semi quantitative characterisation of intracellular distribution of GSK2292767 within lung resident cells, binding and lysosomal uptake and retention.

Unfortunately, this binding and lysosomal work failed during preliminary investigation and so only the imaging of the cell for drug will be investigated, though it is uncertain whether the compound ionises sufficiently to allow detection.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the safety and tolerability of single and repeat doses of GSK2292767 as a dry powder in healthy cigarette smokers. | Safety and tolerability of GSK2292767 as assessed by clinical monitoring of: • Vital Signs • Spirometry • ECG • Laboratory safety data • Adverse events (AEs) |
| Secondary Objectives | Secondary Endpoints |
| To determine the pharmacokinetic profile of single and repeat doses of GSK2292767 as a dry powder in healthy cigarette smokers | <ul> <li>GSK2292767 plasma concentration data and derived pharmacokinetic parameters including area under the plasma drug concentration versus time curve (AUC<sub>(0-t)</sub>, AUC<sub>(0-24)</sub>, AUC<sub>(0-∞)</sub>), maximum observed plasma drug concentration (C<sub>max</sub>), time to maximum observed plasma drug concentration (T<sub>max</sub>),terminal half-life (T<sub>1/2</sub>) and trough concentrations (Cτ) following single and repeated dry powder doses, where data allow.</li> </ul> |
| To investigate the steady-state trough concentration of GSK2292767 in lung epithelial lining fluid (ELF) and Bronchoalveolar lavage (BAL) cell pellet after repeat inhaled dry powder administration in healthy cigarette smokers. | BAL concentrations of GSK2292767 and derived lung ELF and cell pellet deposition parameters. |

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To determine the pharmacodynamic effect of GSK2292767 on the biomarker Phosphatidylinositol (3,4,5)-trisphosphate (PIP3) in induced sputum after single and repeat doses of GSK2292767 administered as a dry powder in healthy cigarette smokers. | PIP3 peak area as a proportion of (PIP3 peak area + Phosphatidylinositol (4,5)-bisphosphate [PIP2] peak area) in induced sputum cells. |
| To explore the intracellular distribution, binding and lysosomal disposition of GSK2292767 from lung resident cells derived from bronchoalveolar lavage at steady-state following repeat administration | Semi quantitative characterisation of intracellular distribution of GSK2292767 within lung resident cells, binding and lysosomal uptake and retention. |
| To generate samples that will be used to characterise the metabolic profile of GSK2292767 in plasma, following single and repeat doses of GSK2292767 administered as a dry powder in healthy cigarette smokers. | Characterisation and quantification of metabolites in plasma. |
| <ul> <li>To collect urine samples only at the<br/>highest proposed dose level to<br/>characterise the renal excretion of<br/>systemically available drug following<br/>inhaled delivery.</li> </ul> | Semi-quantitative characterisation of amount of parent GSK2292767 excreted in urine |

#### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No formal statistical analysis is planned.

A review of preliminary safety and pharmacokinetic data will be conducted prior to selection of the doses for Part A and before confirmation of the dose for Part B. Safety data will be provided by the site at the end of each dosing session. Pharmacokinetic data will be provided by or under the auspices of Clinical Pharmacokinetics Modelling & Simulation (CPMS) using Phoenix WinNonlin.

The decision to proceed to the next dose level of GSK2292767 in Part A and the selection of the daily dose level to be tested in Part B will be made by the GSK Study Team and the investigator based on blinded safety data (AE, vital signs, ECG and laboratory safety test) and preliminary blinded PK data (up to 24 h) obtained in at least 5 subjects on active

drug at the previous dose level. For a detailed description of the dose justification please refer to protocol Section 10.3.4.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects from both study parts have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | <ul> <li>Comprise of all subjects who were<br/>screened</li> </ul> | Listings |
| Safety | <ul> <li>Comprise of all subjects who receive at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | <ul><li>Study Population</li><li>Safety</li><li>Pharmacodynamic</li></ul> |
| Pharmacokinetic | <ul> <li>Subjects in the 'Safety' population for whom a pharmacokinetic sample was obtained and analysed.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | • PK |

#### NOTES:

Please refer to Appendix 11: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| Section 10.1 | Appendix 1: Time & Events |
| Section 10.2 | Appendix 2: Assessment Windows |
| Section 10.3 | Appendix 3: Treatment States and Phases |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| Section 10.7 | Appendix 7: Values of Potential Clinical Importance |
| Section 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses. |
| Section 10.9 | Appendix 9: Population Pharmacokinetic Analyses |
| Section 10.10 | Appendix 10: Abbreviations and Trademarks |
| Section 10.11 | Appendix 11: List of Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gen | erated |
|---|---|---|---|
| | Figure | Table | Listing |
| Randomisation | <u>.</u> | | |
| Randomisation | | | Υ |
| Subject Disposition | | | |
| Subject Disposition | | Υ | |
| Reasons for Screening Failures | | | Υ |
| Important Protocol Deviations | | Υ | Υ |
| Inclusion and Exclusion Criteria Deviations | | Υ | Υ |
| Demography | | | |
| Demographics Characteristics | | Υ | Υ |
| Race & Racial Combinations | | Υ | Υ |
| Study Populations | | Υ | Υ |
| Medical Condition & Concomitant Medications | • | | • |
| Medical Conditions (Current/Past) | | Υ | |
| Concomitant Medication | | Y | |

#### NOTES:

• Y = Yes display generated.

# 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Safety Analyses

#### 7.1.1. Overview of Planned Safety Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

# 7.1.2. During the Study

As required, ongoing data reviews will be conducted by the study team of the unblinded safety data, throughout the trial progression.

#### 7.1.2.1. Dose Escalations

• The principal investigator and medical monitor will provide an overall summary of the required safety data for the dose escalation review for progressing to the next cohort, as defined in the protocol.

# 7.1.3. Final Safety Data

Table 3 provides an overview of the planned safety analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 3 Overview of Planned Safety Analyses

| Endpoint / Parameter/ | Abso | lute | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Display Type | Sum | mary | Indiv | /idual | Sum | mary | Indiv | idual |
| | Т | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | |
| Extent of Exposure | Υ | | | Υ | | | | |
| Adverse Events | | | | | | | | |
| All AEs (Safety population) | Υ | | | Υ | | | | |
| Drug-related AEs | Υ | | | | | | | |
| Serious AEs | | | | Υ | | | | |
| AEs leading to withdrawal | | | | Υ | | | | |
| Relationship between SOC | | | | Υ | | | | |
| and verbatim text | | | | | | | | |
| AEs by Preferred Term | Υ | | | | | | | |
| with Occurrences >=5% in | | | | | | | | |
| any treatment arm | | | | | | | | |
| Laboratory Data | | | | | | | | T |
| Clinical Chemistry | | | | Y1 | Υ | | | |
| Haematology | | | | Υ1 | Y | | | |
| Urinalysis Data | | | | Υ1 | Υ | | | |
| ECG | | | | | | | | |
| ECG Values | | Υ | Υ | Y2 | Υ | | | |
| ECG Findings | Υ | | | Υ | | | | |
| Frequency of Maximum ECG | Υ | | | | | | | |
| Values | | | | | | | | |
| by Pre-Specified Categories | | | | | | | | |
| Vital Signs | | | | | | | | |
| Vital Signs Values | | | | <b>Y</b> 3 | Υ | | | |
| Spirometry | | | | | | | | |
| Lung Function | | | | Υ | Υ | | | |
| Parameters | | | | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1]Two Listings of chemistry and haematology data will be produced. One will list all abnormalities of PCI and the other will list all chemistry/haematology data for all subjects with any chemistry/haematology abnormalities.
- [2]Two listings of ECG data will be produced. One will list all ECG abnormalities of PCI and the other will list all ECG data for all subjects with any ECG PCI values.
- [3]Two listings of vital signs data will be produced. One will list all vital signs abnormalities of PCI and the other will list all vital signs data for all subjects with any vital signs PCI values.

#### 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Pharmacokinetic Analyses

# 8.1.1. Overview of Planned Pharmacokinetic Analyses

The following PK analyses will only be performed if sufficient data are available (i.e., if subjects have well defined plasma profiles). Analyses will be performed on the Pharmacokinetic Population.

#### 8.1.2. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3 Reporting Process & Standards).

# 8.1.2.1. Overview of Planned Pharmacokinetic Analyses for Drug Concentrations

Table 4 provides an overview of the planned pharmacokinetic analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 4 Overview of Planned Pharmacokinetic Data

| Endpoints | | Untrans | sformed | | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indiv | idual | Sum | mary | Individual | |
| | F T | | F | L | F | T | F | L |
| Plasma Drug Concentrations | Υ [1] [2] | Υ | Y [1] | Υ | | Υ | Υ | |
| Derived PK Parameters | | Υ | | Υ | | Υ | | |
| Urine PK Data | | Υ | | | | | | |
| Lung ELF and Cell Pellet | Υ | Υ | | | | | Υ | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Median plots will be generated.

#### 8.1.3. Pharmacokinetic Parameters

### 8.1.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Nonlin Pro.
- All calculations of non-compartmental parameters will be based on actual sampling times recorded during the study.

• Pharmacokinetic parameters described in Table 5 will be determined from plasma GSK2292767 concentration-time data, as data permit.

 Table 5
 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-24) | Area under the concentration-time curve over the dosing interval. |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated as follows: AUC = $AUC(0-t) + C(t)/\lambda z$ . |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Сτ | Trough concentration |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| T½ | Apparent terminal half-life will be calculated as: |
| | t½ = In2 / Lambda_z |
| | (NOTE: λz is the terminal phase rate constant). |

**NOTES:** Additional parameters may be included as required.

#### 8.1.4. BAL Parameters

No pharmacokinetic parameters will be derived for BAL data. The corrected concentrations will be listed, summarised and plotted.

#### 8.1.5. Single Dose Escalation (Part A)

Table 6 Overview of Dose Proportionality Summaries

| Endpoint / Parameter/ | | | Untr | ransfo | rmed | | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stats Analysis | | | Sum | Stat | s Ana | lysis | Summary | | Individual | | | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Dose Proportionality | | | | | | | | | | | | | | |
| Dose Proportionality: | | | | | | | | Υ | | | | | | |
| Power Model | | | | | | | | | | | | | | |
| Dose Proportionality: | | | | | | | | Υ | Υ | | | Υ | | |
| ANOVA Method | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

Boxplots of dose-normalised AUC(0-t), Ctau and Cmax versus dose will be produced, a separate plot for each PK parameter. To calculate the dose normalised parameters, the derived parameter for each dose will be divided by the relevant dose and multiplied by the chosen nominal dose (100ug). If, in the opinion of the Clinical Pharmacology representative, there are a high number of LLQ values at the 100ug dose then another nominal dose will be agreed prior to DBF.

#### 8.1.5.1. Statistical Analysis of Dose Proportionality

The following pharmacokinetic statistical analyses will only be performed if sufficient data are available (i.e. if more than 6 subjects have well defined plasma profiles). If the dose with limited data is at the lower end of the dose range, the data will be excluded and the appropriate analysis conducted on the rest of the data. However if there are non-calculable PK parameter data at intermittent doses no statistical analyses will be performed. A minimum of 3 doses will be required to assess dose proportionality. The assessment of dose proportionality will utilise Part A data only.

# Pharmacokinetic Statistical Analyses for Dose Proportionality: Power Method Endpoint(s)

- AUC(0-t), Cτ, Cmax
- Each endpoint to be assessed separately.

#### **Model Specification**

loge(Y) = β × loge(dose) + loge(α)
 where Y is the pharmacokinetic parameter and loge(α) is an intercept term.

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- The coefficient of the slope with 90% confidence intervals, on the log scale, will be calculated, using the pooled estimate of variance, and used to assess dose proportionality.
- Point estimates and confidence intervals for the slope will be reported to 2 decimal places

The ANOVA method will also be used to assess dose proportionality.

# Pharmacokinetic Statistical Analyses for Dose Proportionality: ANOVA Method Endpoint(s)

- AUC(0-t), Cτ, Cmax
- Each endpoint to be assessed separately.

#### **Model Specification**

- The PK parameter will be dose-normalised prior to loge-transformation by multiplying by reference dose / dose
- Dose will be fitted as a fixed effect, subject as a random effect using DDFM=KR.
- Separate lines will be fitted for each cohort by including terms for cohort and cohort\*log<sub>e</sub>(dose).
   If the slopes are not significantly (p-value<0.05) different from each other, the interaction term will be removed and a single slope estimate obtained. If the slopes are significantly different from each other, a separate slope estimate and associated 90% confidence interval will be reported for each cohort.</p>
- The reference dose will be chosen based on the lowest clinically relevant dose over which PK
  can be adequately described, with each other dose as the test doses in the construction of the
  ratio µ(test)/µ(reference).

# **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Point estimates for the adjusted means on the log<sub>e</sub> scale, the mean difference between each
  dose (test) and the reference dose and associated 90% confidence interval will be constructed
  using the residual variance. These will not be presented.
- The point estimate and confidence interval will then be exponentially back-transformed to allow the presentation of the adjusted (least square) geometric means for each treatment (dose), and point estimates and associated 90% confidence intervals for the ratio test/reference.
- Point estimates and 90% confidence intervals for AUC, Cmax and  $C_{\tau}$  will be reported to 2 decimal places Treatment ratios and 90% Cls will be plotted by dose.
- Plots will also be provided showing the adjusted geometric mean ratio of test to reference treatment (dose) for AUC(0-∞), AUC(0-t), Cτ and Cmax together with 90% confidence interval.

### 8.1.6. Repeat Dose (Part B)

• If more than 1 cohort is recruited in order to investigate more than 1 repeat dose then cohort will be added as a covariate. Only Part B data will be analysed for the repeat dose assessments.

Table 7 Overview of Repeat Dose Summaries

| Endpoint / Parameter/ | | | Unti | ransfo | rmed | | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stats Analysis | | | Summary Individual | | | | Stat | s Ana | lysis | Summary | | Individual | |
| | T | F | Ĺ | T | F | F | Ĺ | Т | F | L | T | F | F | Ĺ |
| Repeat Dose | | | | | | | | | | | | | | |
| Dose Accumulation | | | | | | | | Υ | | | | | | |
| Steady State | | | | | | | | | | | | Υ | | |
| Peak to Trough Ratios | | | | | | | | Υ | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.1.6.1. Statistical Analysis of Dose Accumulation and Steady State

The following pharmacokinetic statistical analyses will only be performed, if sufficient data are available (i.e. if subjects have well defined plasma profiles).

#### **Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

- Dose Accumulation: AUC(0-24), Cτ, Cmax on Day 14 compared to Day 1
- Each endpoint to be assessed separately following a log-transformation.

#### Model Specification

- A mixed effect model will be fitted with day as a fixed effect and subject as a random effect.
- The Kenward & Roger (KR) degrees of freedom approach will be used.
- Day 14 will be compared to Day 1 in order to estimate the accumulation ratio(s)
- The accumulation ratio(s) and 90% confidence interval will be calculated by back-transforming the difference between the least square means for the two days and associated 90% confidence interval.

#### Model Checking & Diagnostics

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Point estimates and confidence intervals for the ratios will be reported to 2 decimal places
- Scatter plots of each endpoint against day will be produced. The data points for each subject
  will be joined with straight lines. If there is more than 1 cohort each treatment will be put on a
  separate page.
- Boxplots of each endpoint against day will be produced. If there is more than 1 cohort each treatment will be put on a separate page.

#### 8.1.6.2. Statistical Analysis of Peak to Trough Ratio

#### **Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

• Peak to trough ratio: Cmax/Ctrough.

# **Model Specification**

- A mixed effect model will be fitted with day\*parameter as a fixed effect and subject as a random effect.
- The Kenward & Roger (KR) degrees of freedom approach will be used.
- Response variable will be the logged peak concentrations and the logged trough concentrations.
- Indicator variables will be included to distinguish between the peak and trough concentration data.
- The differences in Ismeans of the peak and trough concentrations on each day will be back-transformed to obtain estimates of the peak to trough ratios on each day.

# Model Checking & Diagnostics

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 Peak to trough ratios will be tabulated displaying the adjusted mean (and 90% CIs) Cmax and Ctrough values together with the ratios and corresponding 90% CIs.

# 8.1.7. Population Pharmacokinetic Analyses

A PME/MAP compliant file will be generated for this study to enable population PK model development, if possible (dependent on data). Data from subjects from both study parts (Parts A and B) will be provided in this file, even for subjects who may not have received a full dose. Such subjects may be included in any subsequent POP PK analysis.

An example file structure is provided in the attachments in Section 10.11. The PME/MAP compliant file will be produced by or under the auspices of Clinical Statistics (Programming).

# 8.2. Pharmacodynamic Analyses (Parts A and B)

# 8.2.1. Overview of Planned Pharmacodynamic Analyses

Analyses will be performed separately for each study part.

The pharmacodynamic analyses will be based on the Safety population, unless otherwise specified.

Table 8 provides an overview of the planned pharmacodynamic analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

 Table 8
 Overview of Planned Pharmacodynamic Analyses

| Endpoint / | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | | | Untı | ransfo | rmed | | Log-transformed | | | | | | | |
| Туре | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Individual | |
| | Т | F | L | Т | F | F | Г | Т | F | L | Т | F | F | L |
| Phospholipid Data | | | | | | | | | | | | | | |
| PIP2 peak area | | | | Υ | | | Υ | | | | Υ | | Υ | |
| PIP3 peak area | | | | Υ | | | Υ | Υ | Υ | | Υ | | Υ | |
| PIP3 peak area<br>proportion (of PIP2<br>peak area and PIP3<br>peak area) | | | | Υ | | | Υ | Υ | Υ | | Υ | | Υ | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 8.2.2. Planned Pharmacodynamic Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

 PIP3 Peak Area proportion (calculated as a proportion of the sum of PIP2 Peak Area and PIP3 Peak Area i.e. PIP3 Peak Area / (PIP2 Peak Area + PIP3 Peak Area))

#### **Model Specification**

- Repeated measures analysis based on the two replicates for each subject on each study day.
- Replicates are to be modeled using VC (variance components) structure
- Response variable: Loge(PIP3 Peak Area proportion).

The following will be included as fixed effects:

Part A: period, treatment\*daytime

Part B: treatment\*daytime\*base

Where daytime can take the values:

Part A: 'Day 1 3h', 'Day 1 24h'

Part B: 'Baseline', 'Day 1 3h', 'Day 1 24h', 'Day 12 3h', 'Day 12 24h'

Daytime and subject will be fitted as random effects

#### **Model Checking**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Planned Statistical Analyses**

#### **Model Results Presentation**

- Adjusted geometric means for each treatment group will be presented along with 90% confidence intervals (CIs).
- Part A: Point estimates of the treatment differences versus placebo and their associated 90% Cls will be calculated for both timepoints (using the pooled estimate of variance) and back transformed to provide estimates and 90% Cls for the treatment ratios.
- Part B: Point estimates of the daytime differences versus placebo and their associated 90%
   Cls will be calculated (using the pooled estimate of variance) and back transformed to provide estimates and 90% Cls for the treatment ratios at each timepoint.
- Bayesian posterior probabilities of seeing differences from placebo less than 0 (ratio less than 1) will be displayed.
- Adjusted geometric means (for each treatment group and timepoint) and treatment ratios, along with 90% CIs will be plotted.

# 9. REFERENCES

GlaxoSmithKline Document Number 2016N288743\_01 Study ID 202062. A single-centre, double-blind (sponsor open), placebo controlled two part study to evaluate the safety, tolerability and pharmacokinetics of single and repeat doses of GSK2292767 as a dry powder in healthy participants who smoke cigarettes. Report Date 05-Jan-2017.

Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung Volumes and Forced Ventilatory Flows. *Eur Respir J.* 1993;Suppl 16:5-40.

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time and Events |
| Section 10.2 | Appendix 2: Assessment Windows |
| Section 10.3 | Appendix 3: Treatment States & Phases |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | Pharmacokinetic |
| | Pharmacodynamic and or Biomarkers |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.7 | Appendix 7: Values of Potential Clinical Importance |
| Section 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Section 10.9 | Appendix 9: Population Pharmacokinetic Analyses |
| Other RAP App | endices |
| Section 10.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 10.11 | Appendix 11: List of Data Displays |

# 10.1. Appendix 1: Time & Events

# 10.1.1. Protocol Defined Time & Events

# **10.1.1.1. SOA – Part A (Single Dose)**

| | | | Pa | rt A (S | Single | Dose) | Treat | ment | Perio | d | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>-1 | Day 1 (time relative to dosing) | | | | | | | | | | Notes | |
| | Pre dose 0h 5m 30m 45m 1h 2h 3h 4h 6h 8h 12h 24h | | | | | | | | | | | | |
| Admission to Unit | Х | | | | | | | | | | | | |
| Urine Drug/Alcohol breath test | Х | | | | | | | | | | | | |
| Urine Pregnancy test | Х | | | | | | | | | | | | |
| Brief Physical Exam | Х | | | | | | | | | | | Х | |
| Laboratory Assessments | Х | | | | | | | | | | | Х | |
| Meals | Х | | | | | | | | ) | ( | | Х | See Section 6.3.1 of protocol |
| 12-lead ECG (single) | | Х | | | Х | | | | Х | | Х | Х | |
| Vital signs (single) | | Х | | Х | | Х | | | | Х | Х | Х | |

| | | | | Pa | rt A (S | ingle | Dose) | Treat | ment | Perio | d | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>-1 | | | | D | ay 1 ( | time r | elative | to do | sing) | | | | | Notes |
| | | Pre<br>dose | 0h | 5m | 30m | 45m | 1h | 2h | 3h | 4h | 6h | 8h | 12h | 24h | |
| Telemetry | | • | <del>(</del> === | ==== | ==== | :===: | ==== | ==== | ==→ | | | | | | Cardiac telemetry: To start approximately1hr Pre-dose and then continuously for the first 5h post dose. |
| Spirometry (triplicate) | | Х | | | | | Х | | | | | | | | |
| Pharmacokinetic and Metabolite Profile Blood Sample | | Х | | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | |
| Pharmacokinetic Urine Sample | | Х | | ←=== | :===: | ==== | ==== | :===: | ==== | ===→ | | | | | Only for the maximum proposed dose group if escalated up to (2000 µg). |
| Inhaler Training | Х | | | | | | | | | | | | | | |
| Dosing | | | Х | | | | | | | | | | | | |
| Sputum induction | | | | | | | | | Х | | | | | Х | |
| Adverse Event Review | | | <b>←=======→</b> | | | | | | | | | | | | |
| Concomitant Medication Review | | | <b>←=======</b> → | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | Χ | |

# 10.1.1.2. SOA – Part B (Repeat Dose)

| | | | | | | | | Part | B (Re | oeat D | ose) S | tudy D | ay | | | | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | D -2 or<br>D -1 | D1 | D2 | D3 | D4 | D5 | D6 | D7 | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15<br>(D14<br>+24h) | D16<br>(D14<br>+48h | D17<br>(D14<br>+72h | D18<br>(D14<br>+96h | |
| Admission to Unit | Х | | | | | | | | | | | | | | | | | | | |
| Urine Drug/Alcohol | Х | | | | | | | | | | | | | | | | | | | |
| Urine Pregnancy test | Х | | | | | | | | | | | | | | | | | | | |
| Brief Physical Exam | Х | | | | | | | | | | | | | | | | | | | |
| Laboratory Assessments | Х | | X <sup>1</sup> | | X <sup>1</sup> | | X <sup>1</sup> | | X <sup>1</sup> | | X <sup>1</sup> | | X <sup>1</sup> | | X <sup>1</sup> | Х | | | | Perform assessment pre dose |
| Meals | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Х | Х | Χ | Χ | | | | See Section 6.3.1 of protocol |
| 12-lead ECG (single) | х | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | X | | | | 2. Perform assessments pre dose and at 30 mins post dose. |
| Vital signs (single) | Х | <b>X</b> 3 | X <sup>3</sup> | <b>X</b> 3 | <b>X</b> 3 | <b>X</b> 3 | X3 | <b>X</b> 3 | <b>X</b> 3 | X <sup>3</sup> | <b>X</b> 3 | <b>X</b> <sup>3</sup> | <b>X</b> 3 | <b>X</b> 3 | <b>X</b> <sup>3</sup> | Х | | | | 3. Perform assessments pre dose. |
| Spirometry (triplicate) | х | X <sup>4</sup> | X4 | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X4 | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | | | | | 4. Perform assessment pre dose and 1h post dose. |
| Pharmacokinetic Blood<br>Sample | | X <sub>6</sub> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sub>6</sub> | X | X <sup>7</sup> | <b>X</b> <sup>7</sup> | X <sup>7</sup> | 5. pre-dose and 5<br>min post dose.<br>6. pre-dose, 5 mins,<br>30 mins, 45 mins, 1,<br>2, 3, 4, 6, 8 and 12h<br>post dose<br>7. If following Single<br>dose (SD) PK<br>analysis deemed<br>necessary. |

| | | Part B (Repeat Dose) Study Day | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | D -2 or<br>D -1 | D1 | D2 | D3 | D4 | D5 | D6 | D7 | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15<br>(D14<br>+24h) | D16<br>(D14<br>+48h | D17<br>(D14<br>+72h | D18<br>(D14<br>+96h | Notes |
| Blood Sample for<br>Metabolic Profiling | | | | | | | | | | | | | | | X6 | Χ | X <sup>7</sup> | <b>X</b> <sup>7</sup> | <b>X</b> <sup>7</sup> | |
| Urea Blood Sample | | | | | | | | | | | | | | | | Χ | | | | Collect sample just before bronchoscopy |
| Inhaler Training | Χ | | | | | | | | | | | | | | | | | | | , , |
| Dosing | | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | | | | |
| Sputum induction | X11 | X8 | | | | | | | | | | | X <sup>9</sup><br>10 | | | | | | | 8. 3h post dose 9. 3h and 24h 10. Should sputum induction fail or be insufficient at any time point then the participant will be allowed to return 24h later for a further attempt to obtain an adequate sample 11. Should sputum induction fail or be insufficient then the participant will be allowed to return 24h later for a further attempt to obtain an adequate sample. Failure to produce a baseline sample will result in participant withdrawal. |

# CONFIDENTIAL

| | | Part B (Repeat Dose) Study Day | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | D -2 or<br>D -1 | | | D3 | D4 | D5 | D6 | D7 | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15<br>(D14<br>+24h) | D16<br>(D14<br>+48h | D17<br>(D14<br>+72h | D18<br>(D14<br>+96h | Notes |
| Bronchoscopy | | | | | | | | | | | | | | | | Х | | | | |
| Adverse Event Review | | | <b>←=======</b> <del>→</del> | | | | | | | | | | | | | | | | | |
| Concomitant Medication Review | | | ←======→ | | | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | Х | | | | |

# 10.2. Appendix 2: Assessment Windows

# 10.2.1. Definitions of Assessment Windows for Analyses

| Analysis Set / | Parameter | Target | Analysis | Window | Analysis |
|---|---|---|---|---|---|
| Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| e.g. "Safety",<br>"Efficacy" or list<br>specific domains if<br>required | e.g. "All" or list<br>specific<br>parameters<br>(i.e. tests) if<br>required | The target or most desired relative day or relative time value for a given visit. e.g. "Day 7" | e.g. "Day 1" | e.g. "Day<br>10" | e.g. VISIT 1 |
| Pharmacodynamic | Sputum PIP data | Day -2 or Day -1 (Part<br>B) | Predose | | PREDOSE |
| | | Day 1 3h (Parts A and B) | Day 1<br>2h45m | Day 1<br>3h15m | Day 1 3h |
| | | Day 1 24h (Part A) | Day 1<br>22h30m | Day 1<br>25h30m | Day 1 24h |
| | | Day12 3h (Part B) | Day 12 <sup>1</sup><br>2h45m | Day 12 <sup>1</sup><br>3h15m | Day 12 3h |
| | | Day 12 24h (Part B) | Day 12 <sup>1</sup><br>22h30m | Day 12 <sup>1</sup><br>25h30m | Day 12 24h |

#### NOTES:

<sup>•</sup> All other data will be summarised using the planned timepoint.

<sup>[1]</sup> Note that if subject is unable to provide a sputum sample on Day 12, then they may have another attempt on Day 13. If this happens then the Day 12 windowing timing will be relative to the Day 13 dose rather than the Day 12 dose.

# 10.3. Appendix 3: Treatment States and Phases

#### 10.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment unless otherwise specified.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

#### 10.3.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 10.3.2.1. Treatment States for Concomitant Medication Data

| <b>Treatment State</b> | Definition |
|---|---|
| Pre-Treatment | Medication End Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date <= Conmed Start Date ≤ Study Treatment Stop Date |
| | Study Treatment Start Date <= Conmed End Date |
| Post-Treatment | ConMed Start Date > Study Treatment Stop Date |

#### NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 10.3.2.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on PIMS OR value is missing. |

#### NOTES:

If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

#### 10.4.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporti | ng |
| Code | Description | Description <sup>[2]</sup> | Order [1] |
| Α | Placebo inhaled single dose | Placebo | 1 |
| В | 50ug GSK2292767 inhaled single dose | 50ug OD | 2 |
| С | Dose Level 2 GSK2292767 inhaled single dose | 100ug OD | 3 |
| D | Dose Level 3 GSK2292767 inhaled single dose | 200ug OD | 4 |
| E | Dose Level 4 GSK2292767 inhaled single dose | 500ug OD | 5 |
| F | Dose Level 5 GSK2292767 inhaled single dose | 1000ug OD | 6 |
| G | Dose Level 6 GSK2292767 inhaled single dose | 2000ug OD | 7 |
| Н | Placebo inhaled repeat dose | Placebo | 1 |
| I | Dose Level 7 GSK2292767 inhaled repeat dose | XXXXug OD | 2 |

#### NOTES:

- 1. Order represents treatments being presented in TFL, as appropriate.
- 2. Replace X's with the actual agreed dose for the cohort and period.

#### 10.4.2. Baseline Definition & Derivations

#### 10.4.2.1. Baseline Definitions

For all endpoints the baseline value will be the latest pre-dose assessment. For Part A, baseline definitions are applicable to each period. Note that no baseline sputum assessments are planned for Part A so any comparisons will be purely versus placebo at the corresponding timepoints.

#### 10.4.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.4.2. Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

# 10.4.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently supported versions of SAS software (Version 9.4) will be used. | |
| Reporting Area | Reporting Area |
| HARP Server | :: UK1SALX00175.corpnet2.com |
| HARP Area | Two reporting efforts will be set up for this study, 1 for Part A (Final_01) and 1 for Part B (Final_02). |
| QC Spreadsheet | : ARPROD\ GSK 2292767 \202062\Final\Documents |
| <b>Analysis Datasets</b> | |
| Analysis datasets will be created according to Integrated Data Standards Library. | |
| Generation of RTF Files | |
| RTF files will be | generated for all tables |

#### Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Reporting Standards**

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

Continuous Data

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Descriptive | Summary | y Statistics |
|-------------|---------|--------------|
|-------------|---------|--------------|

| Reporting of Pharmacokinetic Concentration Data | |
|---|---|
| Categorical Data | N, n, frequency, % |
| Continuous Data | Trefer to 1002 Statistical Fillicipie 6.66.1 |

| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
|---|---|
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |

Refer to IDSI Statistical Principle 6.06.1

| Reporting of Pharmacokinetic Parameters | |
|---|---|
| Descriptive<br>Summary Statistics<br>(Log Transformed) | <ul> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between and or within geometric coefficient of variation (CVb/w (%)) will be reported.</li> <li>[1] CV<sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data)</li> <li>[2] CV<sub>w</sub> (%) = √ (exp(MSE) - 1) * 100 (MSE = mean square error from mixed effect model of loge-transformed data).</li> </ul> |
| Parameters Not<br>Being Log<br>Transformed | Tmax |
| Summary Tables | All provided PK parameters will be summarised except Lamz, lamzUL, LamzLL, LamzNP and AUC % extrapolated area (if calculated). |
| Listings | Additionally, include the first point, last point and number of points used in the determination of lambda_z for listings. |

#### **Graphical Displays**

- Refer to IDSL Statistical Principles 7.01 to 7.13.
- All graphics will be done using the SGPLOT/SGPANEL/SG template procedures.
- Where possible, n's will be displayed in summary plots.

# 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from randomisation date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### **Insert as Required**

Insert as Required

### 10.5.2. Study Population

# **Demographics**

#### Age

- Age will be calculated based on year of birth compared to the date of the screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / (Height (m))<sup>2</sup>

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### 10.5.3. Safety

#### **ECG Parameters**

#### **RR** Interval

• IF RR interval (msec) is not provided directly, then RR can be derived as:

If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Adverse Events**

#### **AE'S OF Special Interest**

 No AE's of special interest have been defined yet. These will not be identified or summarised for SAC.

# **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

#### 10.5.4. Calculation of Spirometry Screening Parameters

• Derived parameters for spirometry data at screening will be calculated as follows:

#### Predicted Normal FEV<sub>1</sub>

• Predicted Normal FEV<sub>1</sub> will be calculated using the working party of the European Community for Coal and Steel (ECCS) formula [Quanjer, 1993]:

$$\frac{Predicted}{Normal\ FEV1} = b_o * Height + b_1 * Age(Yr) + b_2$$

• The coefficients for male and female subjects are shown in Table 9. Note that no race corrections will be made.

Table 9 Predicted Normal FEV<sub>1</sub> Equation: Coefficients for Male and Female Subjects

| | Height (b₀) | Age (b <sub>1</sub> ) | Intercept (b <sub>2</sub> ) |
|--------|-------------|-----------------------|-----------------------------|
| Male | 0.0430 | -0.029 | -2.49 |
| Female | 0.0395 | -0.025 | -2.60 |

#### % Predicted Normal FEV<sub>1</sub>

$$\frac{\%Predicted}{Normal\ FEV_{1}} = \frac{MaxFEV_{1}}{Predicted\ Normal\ FEV_{1}} *100$$

#### 10.5.5. Pharmacodynamic

#### **Sputum Data**

#### **PIP3 Ratio**

- PIP3 is the analyte of primary interest for the phospholipid data in sputum, and Peak Area data from the mass spectrometer is the endpoint of interest. However, it is acknowledged that there will be some degree of variability between sputum samples due to differences in cell counts, and therefore it is favoured to first normalise PIP3 Peak Area values by (PIP2 Peak Area + PIP3 Peak Area); prior to analysis.
- More specifically the parameter of interest is: PIP3 Peak Area proportion (calculated as a proportion of the sum of PIP2 Peak Area and PIP3 Peak Area i.e. PIP3 Peak Area / (PIP2 Peak Area + PIP3 Peak Area)).
- PIP3 Peak Area, as a proportion of PIP2 Peak Area and PIP3 Peak Area, will be used to calculate the PIP3 Peak Area proportion as follows:

#### **Sputum Data**

$$PIP3$$
  $Peak$   $Area$   $proportion = \frac{PIP3\ Peak\ Area}{PIP2\ Peak\ Area} + PIP3\ Peak\ Area$ 

• PIP3 peak area, (PIP3) may be standardised by dividing by a PIP3 standard e.g. ISDPIP3. Similarly, PIP2 peak area (PIP2) may be standardised by dividing by a PIP2 standard e.g. D6PIP2. Multiple standards will be included in the PIP dataset. The unstandardised PIP2 and PIP3 peak areas will be used in the derivation of the PIP3 peak area proportion for the SAC outputs. However, the choice of standards to be used in the analysis may be explored e.g. through comparison of distributions, linear regression post SAC.

#### 10.5.6. Derivation of BAL/ELF Drug Concentration Data

• Urea concentration data will be used to calculate the dilution effect of the lavage which is used to extract the epithelial lining fluid (ELF) from the lung. A correction for dilution will be applied to all BAL fluid drug concentrations for each wash as follows:

$$ELF\ Drug\ Concentration\ (pg/mL) = \frac{BAL\ Fluid}{Drug\ Concentration} (pg/mL) \times Dilution\ Factor$$

where

$$Dilution \; Factor = \frac{Plasma \; Urea_{pre-bronch}}{BAL \; Urea}$$

• Additionally, for each wash, the Volume of ELF in BAL fluid and the Total Drug in BAL fluid will be calculated as follows:

 $Volume\ of\ ELF\ in\ BAL\ Fluid\ (mL) = BAL\ Fluid\ Volume\ (mL)/Dilution\ Factor$ 

$$Drug \ in \ BAL \ Fluid \ (pg) = \frac{BAL \ Fluid}{Drug \ Concentration} (pg/mL) \times BAL \ Fluid \ Volume \ (mL)$$

• Data will then be pooled across all three washes as follows:
$$Pooled \; ELF \; Drug \; Concentration \; (pg/mL) = \frac{Total \; Drug \; in \; BAL \; Fluid \; (pg)}{Total \; Volume \; of \; ELF \; in \; BAL \; Fluid \; (mL)}$$

### 10.5.7. Derivation of BAL Cell Pellet Drug Concentration Data

• Cell pellet samples are diluted in a 1:5 ratio. Concentrations will be corrected for the dilution before the ratio is calculated on an individual subject level between the raw lavage result for wash 2 and the cell pellet concentration:

Derived cell pellet concentration

- $= \frac{\text{cell pellet concentration x 5}}{\text{wash 2 lavage concentration}} \text{ x derived pooled lavage ELF concentration}$
- Only the derived concentrations will be included in the listing.

# 10.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

## 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as the completion of all phases of the study including the follow up visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table. Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| PK and PD | <ul> <li>It is possible that not enough data points will be captured for the sputum at baseline (Part B) and/or at a specific post dose time point for all treatment groups. In such a situation, data should only be listed. No attempt should be made to summarise or statistically analyse the data.</li> <li>The decision for the summary/statistical analysis of PK and PD data should be made once the study team and statistician have reviewed the totality of available data.</li> <li>Any values below the Lower Limit of Quantification (LLQ) will be assigned a value of ½ LLQ for display purposes in Figures and for computation of summary statistics. Any values above the Upper Limit of Quantification (ULQ) will be assigned to the ULQ for display purposes in Figures and for computation of summary statistics. If multiple LLQ and /or ULQ values are available per assay (for example if multiple runs with different standard curves are utilised) then the LLQ and/or ULQ value used for the above imputation shall be the minimum of the available LLQs and/or the maximum of the ULQs. Where biomarker concentrations are from an assay of an increased dilution factor the LLQ and ULQ will be multiplied by this factor.</li> <li>If the number of LLQ (and/or ULQ) values is large for an Individual biomarker then alternative analysis methods such as TOBIT analysis may be required. "Large" is hard to define prospectively and may depend upon the dataset in</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | question. Any such methodology will be documented in the statistical contributions to the study report. |
| | <ul> <li>Imputed values will be used in tables and figures, unless the proportion of<br/>imputed values at a given time point is large, in which case the summary<br/>statistics may not be presented for that time point and/or alternative actions will<br/>be taken and documented in the study report.</li> </ul> |
| | <ul> <li>Where values are imputed, the number of such imputations will be included as a<br/>summary statistic in the relevant summary tables.</li> </ul> |

### 10.6.2.1. Handling of Missing Dates

PIMS does not capture partial dates, all AEs and con meds will have full dates. Prior medications will have duration and full stop date.

## 10.6.2.2. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|----------------|----------------------------------|
| PK and PD data | Missing data will not be imputed |

# 10.7. Appendix 7: Values of Potential Clinical Importance

## 10.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | D :: ( | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| | • | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 8.0 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 10.7.2. ECG

| ECG Parameter | Units | Clinical Cor | ncern Range |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | > 450 <sup>1</sup> | |
| Absolute PR Interval | msec | < 110 <sup>1</sup> | > 220 ¹ |
| Absolute QRS Interval | msec | < 75 <sup>1</sup> | > 110 ¹ |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 60 ¹ | |

NOTES: 1 Represent standard ECG values of PCI for HV studies

## 10.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### 10.8.1. Statistical Analysis Assumptions

| Endpoint(s) | • | Dose proportionality, accumulation, peak to trough ratio, PIP3 Ratio |
|---|---|---|
| Analysis | • | Mixed effects models |

- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

## 10.9. Appendix 9: Population Pharmacokinetic Analyses

#### 10.9.1. POP PK Dataset creation

A POP PK analysis compliant dataset will be created using the following example structure.

The PME/MAP compliant file structure is a space-delimited file with each row containing the following columns of information.

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| STUD | Protocol Number | Varchar | - | 202062 |
| SUBJ | Subject identifier in study | Varchar | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Varchar | - | |
| LABL | Indicator field describing the type of assessment in that record | Varchar | | LABL=DOSE for a dosing event and LABL=CONC for a concentration event |
| AMT | Dose | Decimal | Mcg | |
| TMT | Treatment Identifier | Integer | - | TMT = 0 for placebo and AMT for dose levels |
| VISIT | Study visit | Integer | - | Maximum 10 characters (numeric or text). |
| DAY | Study day | Integer | - | numeric , Actual Study Day Number |
| DATETIME | Date and time of<br>Dose or<br>measurement | YYYY-MM-<br>DD<br>HH:MM:SS | - | Date and time of assessment. The supported range is '1000-01-01 00:00:00' to '9999-12-31 23:59:59' |
| TIME | Actual time relative to first active dose | Decimal | Hours | Hours since first active dose. |
| RTLD | Actual time relative to last active dose | Decimal | Hours | When LABL = DOSE, RTLD = 0 Hours since last active dose. For predose sample. For predose sample, TIME is relative to previous morning (am) dose on previous Day X |
| CONC | Value of the variable captured in the LABL/TIME pair | Decimal<br>(12,4) | As detailed for variable below | |
| EVID | Event ID | Integer | | EVID=1 for a dosing event record (where AMT is also positive number) and EVID=0 otherwise (where AMT is 0) |
| MDV | Missing Data<br>Variable | Integer | - | MDV=1 when EVID=1 and MDV=0 when EVID=0 |
| NQ | Non Quantifiable<br>Data | Integer | | If CONC is NQ then NQ=1 else 0 |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| IND | BQL indicator | Integer | - | If CONC is NQ then IND=1, else IND=0 |
| LLQ | Lower Limit of quantification | Integer | pg/mL | Lower limit of quantification for specific analyte |
| II | Interdose interval | Decimal | Hours | Interdose Interval (II) gives the time between doses (24 h for once daily dosing). Il should be a positive number if and only if the AMT data item is a positive number and has the same units as the TIME data item. For CONC records, II should be zero. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| SEXTXT | Subject gender | Varchar | - | MALE (male) or FEMALE (female) |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| TOBAC | Tobacco Use | Decimal | | Number of pack years (=number of cigarettes per day/20))X number years smoked |

## **Example Dataset**

| D | SUBJ | CENT | STUD | LABL | AMT | TMT | VISIT | DAY | DATETIME | TIME | RTLD | CONC | EVID | MDV | NQ | IND | LLQ | = |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 2 | 1 | PPD<br>1:06:12:00 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | |
| | | | DB21<br>13361 | DOSE_UM<br>_361_MO | 1<br>2<br>5 | 3 | 2 | 1 | PPD<br>1:06:39:00 | 0 | 0 | | 1 | 1 | 0 | 0 | | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 2 | 1 | PPD<br>1:06:44:00 | 0.0 | 0.<br>08 | 11<br>7.<br>2 | 0 | 0 | 0 | 0 | 1 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 2 | 1 | PPD<br>1:07:00:00 | 0.3<br>5 | 0.<br>35 | 84<br>.4 | 0 | 0 | 0 | 0 | 1 0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 2 | 1 | PPD<br>1:15:16:00 | 8.6<br>2 | 8.<br>62 | 25<br>.5 | 0 | 0 | 0 | 0 | 1 0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 2 | 2 | PPD<br>1:05:40:00 | 23.<br>02 | 23<br>.0<br>2 | 0 | 0 | 0 | 1 | 1 | 1 | |

| | | | | | | | | | D | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ₽ | SUBJ | CENT | STUD | LABL | AMT | TMT | VISIT | DAY | DATETIME | TIME | RTLD | CONC | EVID | MDV | NQ | IND | LLQ | = |
| PPD | | | DB21<br>13361 | DOSE_UM<br>_361_MO | 1<br>2<br>5 | 3 | 6 | 8<br>5 | PPD<br>1:07:15:00 | 201<br>6.6 | 0 | | 4 | 1 | 0 | 0 | | 2 |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 6 | 8<br>5 | PPD<br>1:07:17:00 | 201<br>6.6<br>3 | 0.<br>03 | 10<br>9.<br>3 | 0 | 0 | 0 | 0 | 1 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 6 | 8<br>5 | PPD<br>1:07:50:00 | 201<br>7.1<br>8 | 0.<br>58 | 49<br>.8 | 0 | 0 | 0 | 0 | 1<br>0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 6 | 8<br>5 | PPD<br>1:13:17:00 | 202<br>2.6<br>3 | 6.<br>03 | 31<br>.9 | 0 | 0 | 0 | 0 | 1<br>0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 6 | 8<br>5 | PPD<br>1:06:07:00 | 201<br>5.4<br>7 | .8<br>7 | 23<br>.8 | 0 | 0 | 0 | 0 | 1<br>0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 6 | 8 | PPD<br>1:06:23:00 | 203<br>9.7<br>3 | 23<br>.1<br>3 | 25<br>.6 | 0 | 0 | 0 | 0 | 1 | |
| | | | DB21<br>13361 | DOSE_UM<br>_361_MO | 1<br>2<br>5 | 3 | 8 | 1<br>6<br>9 | PPD<br>1:06:54:00 | 403<br>2.2<br>5 | 0 | | 4 | 1 | 0 | 0 | | 2 |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 8 | 1<br>6<br>9 | PPD<br>1:06:56:00 | 403<br>2.2<br>8 | 0.<br>03 | 16<br>8 | 0 | 0 | 0 | 0 | 1 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 8 | 1<br>6<br>9 | PPD<br>1:07:29:00 | 403<br>2.8<br>3 | 0.<br>58 | 29<br>.9 | 0 | 0 | 0 | 0 | 1<br>0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 8 | 1<br>6<br>9 | PPD<br>1:13:00:00 | 403<br>8.3<br>5 | 6.<br>1 | 16<br>.9 | 0 | 0 | 0 | 0 | 1 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 8 | 1<br>6<br>9 | PPD<br>1:06:14:00 | 403<br>1.5<br>8 | 23<br>.2<br>3 | 0 | 0 | 0 | 1 | 1 | 1 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_MO | 0 | 3 | 8 | 1<br>7<br>0 | PPD<br>1:06:48:00 | 405<br>6.1<br>5 | 23<br>.9 | 0 | 0 | 0 | 1 | 1 | 1<br>0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_CO | 0 | 2 | 2 | 1 | PPD<br>1:07:08:00 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | |
| | | | DB21<br>13361 | DOSE_UM<br>_361_CO | 1<br>2<br>5 | 2 | 2 | 1 | PPD<br>1:08:00:00 | 0 | 0 | | 1 | 1 | 0 | 0 | | |
| | | | DB21<br>13361 | CONC_UM<br>_361_CO | 0 | 2 | 2 | 1 | PPD<br>1:08:12:00 | 0.2 | 0.<br>2 | 76<br>.2 | 0 | 0 | 0 | 0 | 1<br>0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_CO | 0 | 2 | 2 | 1 | PPD<br>1:08:23:00 | 0.3<br>8 | 0.<br>38 | 49<br>.6 | 0 | 0 | 0 | 0 | 1<br>0 | |
| | | | DB21<br>13361 | CONC_UM<br>_361_CO | 0 | 2 | 2 | 1 | PPD<br>1:14:00:00 | 6 | 6 | 19<br>.2 | 0 | 0 | 0 | 0 | 1 | |

| | | | | 1 | 1 | |
|-----|-----|-----|--------|------|------|-------|
| AGE | HT | SEX | SEXTXT | WT | BMI | TOBAC |
| 69 | 156 | 2 | F | 48.6 | 20 | 78 |
| 55 | 163 | 2 | F | 86.3 | 32.5 | 40 |
| 55 | 163 | 2 | F | 86.3 | 32.5 | 40 |
| 55 | 163 | 2 | F | 86.3 | 32.5 | 40 |
| 55 | 163 | 2 | F | 86.3 | 32.5 | 40 |
| 55 | 163 | 2 | F | 86.3 | 32.5 | 40 |
| 55 | 163 | 2 | F | 86.3 | 32.5 | 40 |

# 10.10. Appendix 10 – Abbreviations & Trade Marks

# 10.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

### 10.10.2. Trademarks

Trademarks of the GlaxoSmithKline Group of Companies

HARP

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

WinNonlin

## 10.11. Appendix 11: List of Data Displays

## 10.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Safety | 2.1 to 2.n | 2.1 to 2.n |
| Pharmacokinetic | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacodynamic and / or Biomarker | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacokinetic / Pharmacodynamic | 5.1 to 5.n | 5.1 to 5.n |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

#### 10.11.2. Deliverable

| Delivery Priority | Description |
|-------------------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

#### NOTES:

• Parts A and B will be reported as part of the same SAC deliverable.

# 10.11.3. Study Population Tables

| Study P | opulation Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Part A ( | Single Dose E | scalation): Subjec | t Disposition | | |
| 1.101 | Screened<br>(Part A) | ES1 | Summary of Subject Disposition (Single Dose) | | SAC |
| 1.102 | Screened<br>(Part A) | ES6 | Summary of Reasons for Screening Failure (Single Dose) | | SAC |
| 1.103 | Safety (Part<br>A) | DV1a | Summary of Important Protocol Deviations (Single Dose) | | SAC |
| 1.104 | Safety (Part<br>A) | DV1a | Summary of All Inclusion/Exclusion Criteria Deviations (Single Dose) | | SAC |
| Part B ( | Repeat Dose): | Subject Dispositi | on | | |
| 1.201 | Screened<br>(Part B) | ES1 | Summary of Subject Disposition (Repeat Dose) | | SAC |
| 1.202 | Screened<br>(Part B) | ES6 | Summary of Reasons for Screening Failure (Repeat Dose) | | SAC |
| 1.203 | Safety (Part<br>B) | DV1a | Summary of Important Protocol Deviations (Repeat Dose) | | SAC |
| 1.204 | Safety (Part<br>B) | DV1a | Summary of All Inclusion/Exclusion Criteria Deviations (Repeat Dose) | | SAC |

| Study P | opulation Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Part A ( | Single Dose Es | scalation): Demog | raphics | | |
| 1.105 | Safety (Part<br>A) | DM1 | Summary of Demographic Characteristics (Single Dose) | Include baseline FEV1 and %predicted normal FEV1. | SAC |
| 1.106 | Safety (Part<br>A) | DM5 | Summary of Race and Racial Combinations (Single Dose) | | SAC |
| 1.107 | Safety (Part<br>A) | SA1 | Summary of Study Populations (Single Dose) | | SAC |
| Part B ( | Part B (Repeat Dose): Demographics | | | | |
| 1.205 | Safety (Part<br>B) | DM1 | Summary of Demographic Characteristics (Repeat Dose) | Include baseline FEV1 and %predicted normal FEV1. | SAC |
| 1.206 | Safety (Part<br>B) | DM5 | Summary of Race and Racial Combinations (Repeat Dose) | | SAC |
| 1.207 | Screened<br>(Part B) | SA1 | Summary of Study Populations (Repeat Dose) | | SAC |
| Part A ( | Single Dose Es | scalation): Medica | l Condition & Con Meds | | |
| 1.108 | Safety (Part<br>A) | MH1 | Summary of Current/Past Medical Conditions (Single Dose) | | SAC |
| 1.109 | Safety (Part<br>A) | CM1 | Summary of Concomitant Medications (Single Dose) | | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Part B ( | Part B (Repeat Dose): Medical Condition & Con Meds | | | | |
| 1.208 | Safety (Part<br>B) | MH1 | Summary of Current/Past Medical Conditions (Repeat Dose) | | SAC |
| 1.209 | Safety (Part<br>B) | CM1 | Summary of Concomitant Medications (Repeat Dose) | | SAC |

# 10.11.4. Safety Tables

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A ( | Single Dose Es | scalation): Exposi | ıre | | |
| 2.101 | Safety (Part<br>A) | EX1 | Summary of Extent of Exposure to Study Treatment (Single Dose) | | SAC |
| Part B ( | Part B (Repeat Dose): Exposure | | | | |
| 2.201 | Safety (Part<br>B) | EX1 | Summary of Extent of Exposure to Study Treatment (Repeat Dose) | | SAC |
| Part A ( | Single Dose Es | scalation): Advers | e Events | | |
| 2.102 | Safety (Part<br>A) | CP_AE1x | Summary of All Adverse Events by System Organ Class (Single Dose) | Include total column. | SAC |
| 2.103 | Safety (Part<br>A) | CP_AE1x | Summary of Drug-Related Adverse Events by System Organ Class (Single Dose) | Include total column. | SAC |

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.104 | Safety (Part<br>A) | AE15/EMA_AE | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences, Single Dose) | | SAC |
| Part B ( | Repeat Dose): | Adverse Events | | 1 | |
| 2.202 | Safety (Part<br>B) | CP_AE1p | Summary of All Adverse Events by System Organ Class (Repeat Dose) | Include total column. | SAC |
| 2.203 | Safety (Part<br>B) | CP_AE1p | Summary of Drug-Related Adverse Events by System Organ Class (Repeat Dose) | Include total column. | SAC |
| 2.204 | Safety (Part<br>B) | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences, Repeat Dose) | | SAC |
| Part A ( | Single Dose Es | scalation): Labs | | ' | |
| 2.105 | Safety (Part<br>A) | LB1 | Summary of Chemistry Changes from Baseline by Visit (Single Dose) | | SAC |
| 2.106 | Safety (Part<br>A) | LB3 | Summary of Emergent Chemistry Results by Potential Clinical Importance Criteria (Single Dose) | | SAC |
| 2.107 | Safety (Part<br>A) | LB1 | Summary of Haematology Changes from Baseline by Visit (Single Dose) | | SAC |
| 2.108 | Safety (Part<br>A) | LB3 | Summary of Emergent Chemistry Results by Potential Clinical Importance Criteria (Single Dose) | | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B ( | (Repeat Dose): | Labs | | | |
| 2.205 | Safety (Part<br>B) | LB1 | Summary of Chemistry Changes from Baseline by Visit (Repeat Dose) | | SAC |
| 2.206 | Safety (Part<br>B) | LB3 | Summary of Emergent Chemistry Results by Potential Clinical Importance Criteria (Repeat Dose) | | SAC |
| 2.207 | Safety (Part<br>B) | LB1 | Summary of Haematology Changes from Baseline by Visit (Repeat Dose) | | SAC |
| 2.208 | Safety (Part<br>B) | LB3 | Summary of Emergent Chemistry Results by Potential Clinical Importance Criteria (Repeat Dose) | | SAC |
| Part A | (Single Dose E | scalation): ECGs | | | |
| 2.109 | Safety (Part<br>A) | EG2 | Summary of Change from Baseline in ECG Values by Visit. (Single Dose) | | SAC |
| 2.110 | Safety (Part<br>A) | EG1 | Summary of Maximum Emergent QTc Values by Category. (Single Dose) | | SAC |
| 2.111 | Safety (Part<br>A) | EG1 | Summary of 12-Lead ECG Findings (Single Dose) | | SAC |
| Part B ( | (Repeat Dose): | ECGs | | | |
| 2.209 | Safety (Part<br>B) | EG2 | Summary of Change from Baseline in ECG Values by Visit. (Repeat Dose) | | SAC |
| 2.210 | Safety (Part<br>B) | EG1 | Summary of Maximum Emergent QTc Values by Category. (Repeat Dose) | | SAC |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.211 | Safety (Part<br>B) | EG1 | Summary of 12-Lead ECG Findings (Single Dose) | | SAC |
| Part A ( | Single Dose Es | scalation): Vital Si | gns | | |
| 2.112 | Safety (Part<br>A) | VS1 | Summary of Change from Baseline in Vital Signs by Visit (Single Dose) | Include the Respiration Rate and Tympanic Temperature | SAC |
| Part B ( | Repeat Dose): | Vital Signs | | | |
| 2.212 | Safety (Part<br>B) | VS1 | Summary of Change from Baseline in Vital Signs by Visit (Repeat Dose) | Include the Respiration Rate and Tympanic Temperature | SAC |
| Part A ( | Single Dose Es | scalation): Spirom | etry | | |
| 2.113 | Safety (Part<br>A) | PD_PFT1 | Summary of Lung Function Data (Single Dose) | | SAC |
| Part B ( | Part B (Repeat Dose): Spirometry | | | | |
| 2.213 | Safety (Part<br>B) | PD_PFT1 | Summary of Lung Function Data (Repeat Dose) | | SAC |

# 10.11.5. Safety Figures

| Safety | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | art A (Single Dose Escalation): ECGs | | | | |
| 2.101 | Safety (Part<br>A) | Fig 2.1 from /arenv/arprod/ gsk2269557/p ii116617/part_ c/drivers/f_qtc _boxplot_part c.sas | Box Plots of QTcF and QTcB Over Time (Single Dose) | One page for each of QTcB and QTcF | SAC |
| Part B | Single Dose E | scalation): ECGs | | | |
| 2.201 | Safety (Part<br>B) | Fig 2.2 from<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/part_<br>b/drivers/f_qtc<br>_boxplot_part<br>b.sas | Box Plots of QTcF and QTcB Over Time (Repeat Dose) | One page for each of QTcB and QTcF | SAC |
| 2.202 | Safety (Part<br>B) | Fig 2.4 from<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/part_<br>b/drivers/f_qtc<br>indiv_partb.sa<br>s | Plot of Individual Subject QTcF and QTcB Over Time (Repeat Dose) | | SAC |

### 10.11.6. Pharmacokinetic Tables

| Pharma | acokinetic : Tal | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | (Single Dose): | Pharmacokinetic ( | Concentrations and Parameters | | |
| 3.101 | PK (Part A) | PKCT1 | Summary of Plasma GSK2292767 Pharmacokinetic Concentration-Time Data (Single Dose) | | SAC |
| 3.102 | PK (Part A) | PKPT1 | Summary of Derived Plasma GSK2292767 Pharmacokinetic Parameters (Single Dose) | Only summarise for AUC(0-t), AUC(0-24), AUC(0-∞), Cmax, Ctau, Tmax, Thalf, Lambda_z. | SAC |
| 3.103 | PK (Part A) | PKPT3 | Summary of Derived Plasma GSK2292767 Pharmacokinetic Parameters (log transformed, Single Dose)) | | SAC |
| 3.104 | PK (Part A) | PKCT1 | Summary of GSK2292767 Pharmacokinetic Urine Excretion Rate-Time Data [units] (Single Dose) | Only for the highest dose. | SAC |
| Part A | (Single Dose): | Dose Proportional | lity | | |
| 3.105 | PK (Part A) | See Table 3.8<br>in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/parts_cb<br>/drivers/t_pkpo<br>wer_partcb.sas | Summary of Results of Statistical Analysis of Plasma<br>GSK2292767 Cmax, AUC(0-t) and Ctau to Assess Dose<br>Proportionality (Single Dose), Power Model | | SAC |
| 3.106 | PK (Part A) | Fig 3.10 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/parts_cb<br>/drivers/t_pkacc<br>um_stat_partcb<br>.sas | Summary of Results of Statistical Analysis of Plasma<br>GSK2292767 Cmax, AUC(0-t) and Ctau to Assess Dose<br>Proportionality (Single Dose), ANOVA Model | | SAC |

| Pharma | acokinetic : Tak | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B | (Repeat Dose): | Pharmacokinetic | Concentrations and Parameters | | |
| 3.201 | PK (Part B) | PKCT1 | Summary of Plasma GSK2292767 Pharmacokinetic Concentration-Time Data (Repeat Dose) | | SAC |
| 3.202 | PK (Part B) | PKPT1 | Summary of Derived Plasma GSK2292767 Pharmacokinetic Parameters (Repeat Dose) | Only summarise for AUC(0-t), AUC(0-24), AUC(0-∞), Cmax, Ctau, Tmax, Thalf, Lambda_z. | SAC |
| 3.203 | PK (Part B) | PKPT3 | Summary of Derived Plasma GSK2292767 Pharmacokinetic Parameters (log transformed) (Repeat Dose) | | SAC |
| Part B | (Repeat Dose) | Statistical Analyse | es | | |
| 3.204 | PK (Part B) | Similar to Table 3.10 in /arenv/arprod/g sk2269557/pii1 16617/parts_cb /drivers/t_pkacc um_stat_partcb .sas | Summary of Statistical Analysis of Plasma GSK2292767 AUC(0-24), Cmax and Ctau Accumulation and Peak: Trough Ratios (Day 14 versus Day 1, Repeat Dose) | Each endpoint to be assessed separately. | SAC |
| Part B | (Repeat Dose): | Lung ELF and Ce | II Pellet Data | | |
| 3.205 | PK (Part B) | See Table<br>11.16 in<br>PII115517/Part<br>_C_Cohort_5 | Summary of Urea Dilution Factor Data (Repeat Dose) | | SAC |
| 3.206 | PK (Part B) | See Table 11.17 in PII115517/Part _C_Cohort_5 | Summary of Derived Lung ELF and Cell Pellet GSK2292767<br>Pharmacokinetic Concentrations and Volume Data (Repeat<br>Dose) | | SAC |

# 10.11.7. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | Single Dose Es | scalation): Pharm | acokinetic Concentrations | | |
| 3.101 | PK (Part A) | PKCF1x | Individual Subject Plasma GSK2292767 Concentration-Time Plots (Linear and Semi-log) by Treatment (Single Dose) | One treatment per page (all subjects within a treatment group on one plot). Add a horizontal line at yaxis = 20 pg/mL and footnote: LLQ = 20 pg/mL,Set pre-dose NQs to missing. | SAC |
| 3.102 | PK (Part A) | PKCF3 | Median Plasma GSK2292767 Concentration-Time Plot (Linear and Semi-Log, Single Dose) | | SAC |
| Part B ( | Repeat Dose): | Pharmacokinetic | Concentrations | | |
| 3.201 | PK (Part B) | PKCF1 | Individual Subject Plasma GSK2292767 Concentration-Time Plots (Linear and Semi-log) by Treatment (Repeat Dose) | If more than one cohort, then 1 cohort per page (all subjects within a treatment group on one plot). Add a horizontal line at y-axis = 20 pg/mL and footnote: LLQ = 20 pg/mL,Set pre-dose NQs to missing. | SAC |
| 3.202 | PK (Part B) | PKCF3 | Median (+ SD) Plasma GSK2292767 Concentration-Time Plot (Linear and Semi-Log, Repeat Dose) | Ĭ | SAC |

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Dose P | roportionality | | | | |
| 3.103 | PK (Part A ) | Fig 3.9 in<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/parts<br>_cb/drivers/f_<br>pkcmax_dose<br>norm_partcb.s<br>as | Box Plot of Dose Normalised Plasma GSK2292767 PK Parameters against Dose (Single Dose) | Separate plots for AUC(0-t), Ctau and Cmax | SAC |
| 3.104 | PK (Part A) | Fig 3.10 from<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/parts<br>_cb/drivers/f_<br>pkanova_part<br>cb.sas | Plot of Adjusted Geometric Mean Treatment Ratios and 90% Cls for Plasma GSK2292767 AUC (0-t) to Assess Plasma Dose Proportionality (Single Dose, ANOVA Model) | | SAC |
| Part B ( | Repeat Dose): | Dose Accumulati | on, Steady State and Peak to Trough Ratios | | |
| 3.203 | PK (Part B) | Fig 3.11 from<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/parts<br>_cb/drivers/f_<br>pkcmax_boxpl<br>ot_partcb.sas | Box Plots of GSK2292767 Plasma PK Parameters by Day (Repeat Dose) | Exclude mean value. Raw means.<br>Cmax, Ctrough and peak to trough<br>ratio on separate pages | SAC |

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B | (Repeat Dose): | Lung ELF and Ce | II Pellet Data | | |
| 3.204 | PK (Part B) | Figure 3.15 in<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/part_<br>b/drivers/fig_3<br>_15_elf.sas | Individual Subject Derived Lung ELF GSK2292767<br>Concentrations Plot (Semi-Log) – Individual Washes (Repeat<br>Dose) | Exclude placebo data. Minor tick marks on x-axis (actual rel time). Initially don't join subjects. Add legend to identify wash no. To be reviewed dependent on data distribution as it may be useful to join lines and plot planned times if the plot doesn't look too messy. | SAC |
| 3.205 | PK (Part B) | Figure 3.16 in<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/part_<br>b/drivers/fig_3<br>_16_elf.sas | Median Plasma and Individual Subject Derived Lung ELF and Cell Pellet GSK2292767 Concentrations Plot (Semi-Log) – Pooled Washes (Repeat Dose) | Exclude placebo data. To only display day 14 data. Minimum y-axis value should be set to 1000 pg/mL Set pre-dose plasma NQs to missing. Legend to identify plasma/ELF and Subjid. Plasma based on planned rel. Time; ELF on actual rel time of Wash 1 Cell Pellet concentration to only be shown for Wash 2 data, ELF data will be the pooled sample. These should be explained within footnote. Jitter these points to the left and right if any of the two sets of points are seen to overlap. | SAC |
| 3.206 | PK (Part B) | Figure 3.17 in<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/part_<br>b/drivers/fig_3<br>_17_pelf.sas | Box Plots of Cell Pellet and Pooled ELF GSK2292767<br>Concentrations (Repeat Dose) | 2 box and whisker plots side by side. Would expect plots to look similar to each other. | SAC |

# 10.11.8. Pharmacodynamic Tables

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A | Single Dose): I | PIP Data | | | |
| 4.101 | Safety (Part<br>A) | See Table 4.4<br>in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/parts_cb<br>/drivers/t_pip_p<br>artcb.sas | Summary of Phospholipid Data in Sputum (Single Dose) | Only include evaluable data and include footnote if any non-evaluable. Summarise geometric mean of reps. Include PIP3 Peak Area, PIP2 Peak Area and PIP3 Peak Area Proportion. | SAC |
| 4.102 | Safety (Part<br>A) | See Table 4.5<br>in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/parts_cb<br>/drivers/t_pip_n<br>ottfrz_stat_part<br>cb.sas | Summary of Results of Statistical Analysis of Phospholipid Data in Sputum (Single Dose) | Include PIP3 Peak Area and PIP3 Peak Area Proportion if appropriate. List PIP3 Peak Area Proportion first if analysed. Add Bayesian posterior probabilities | SAC |

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part B ( | Repeat Dose): | PIP Data | | | |
| 4.201 | Safety (Part<br>B) | See Table 4.4<br>in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/parts_cb<br>/drivers/t_pip_p<br>artcb.sas | Summary of Phospholipid Data in Sputum (Repeat Dose) | Only include evaluable data and include footnote if any non-evaluable. Summarise geometric mean of reps. Include PIP3 Peak Area, PIP2 Peak Area and PIP3 Peak Area Proportion. | SAC |
| 4.202 | Safety (Part<br>B) | See Table 4.5<br>in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/parts_cb<br>/drivers/t_pip_n<br>ottfrz_stat_part<br>cb.sas | Summary of Results of Statistical Analysis of Phospholipid Data in Sputum (Repeat Dose) | Include PIP3 Peak Area and PIP3 Peak Area Proportion if appropriate. List PIP3 Peak Area Proportion first if analysed. Add Bayesian posterior probabilities | SAC |

# 10.11.9. Pharmacodynamic Figures

| Pharma | acodynamic: Fi | gures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part A ( | Single Dose): I | PIP Data | | | |
| 4.101 | Safety (Part<br>A) | Fig 4.23 in /arenv/arprod/ gsk2269557/p ii116617/parts _cb/drivers/f_ pipratio_indiv _partcb.sas | Plot of Individual Subject Phospholipid Data in Sputum by Treatment (Single Dose) | Plot PIP3 peak area, PIP2 peak area and PIP2+PIP3 Peak Areas (geo means of reps) by treatment (x-axis). Include all subjects on one plot. Y-axis: log scale; subject data points to be joined for each analyte. Symbols/colour to identify PIP2 peak area, PIP3 peak area etc. in legend. | SAC |
| 4.102 | Safety (Part<br>A) | Fig 4.8 in /arenv/arprod/ gsk2269557/p ii116617/parts _cb/drivers/f_ pipratio_nottfr z_mean_partc b.sas | Plot of Adjusted Geometric Means and 90% CIs of Phospholipid Data in Sputum (Single Dose) | Y-axis: log scale<br>PIP3 peak area Proportion and<br>PIP3 Peak area | SAC |
| Part B ( | Repeat Dose): | PIP Data | | | |
| 4.201 | Safety (Part<br>B) | Fig 4.4 in<br>/arenv/arprod/<br>gsk2269557/p<br>ii116617/interi<br>m_c/drivers/f_<br>pipratioindiv_<br>partc.sas | Plot of Individual Subject Phospholipid Data in Sputum by Treatment and Time (Repeat Dose) | PIP3 Peak Area Proportion and PIP3 Peak Area | SAC |

| Pharma | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.202 | Safety (Part<br>B) | Fig 4.9 in /arenv/arprod/ gsk2269557/p ii116617/parts _cb/drivers/f_ pipratio_nottfr z_diff_partcb. sas | Plot of Adjusted Treatment Ratios and 90% Cls of Phospholipid Data in Sputum (Repeat Dose) | Y-axis: log scale<br>PIP3 Peak Area Proportion and<br>PIP3 Peak Area | SAC |

# 10.11.10. Pharmacokinetic / Pharmacodynamic Figures

(Note: No PK/PD Summary Tables are planned)

| Pharma | Pharmacokinetic / Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK vs S | Sputum PIP3 R | atio | | | |
| 5.101 | PK (Part A) | Fig 6.2 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>15119/part_b/dr<br>ivers/f_pcon_vs<br>_biom | Scatter Plot of Plasma GSK2292767 Pharmacokinetic Concentration vs PIP3 Peak Area Proportion (Single Dose) | Use different symbols for Day 1 3h and Day 1 24h. | SAC |
| 5.201 | PK (Part B) | Fig 6.2 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>15119/part_b/dr<br>ivers/f_pcon_vs<br>_biom | Scatter Plot of Plasma GSK2292767 Pharmacokinetic Concentration vs PIP3 Peak Area Proportion (Repeat Dose) | Use different symbols for Day 1 3h Day 12 3h and Day 12 24h. | SAC |

# 10.11.11. ICH Listings: Part A (Single Dose Escalation)

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Treatm | ent Information | 1 | | | |
| 1. | Screened<br>(Part A) | CP_TA2 | Listing of Randomised and Actual Treatments (Single Dose) | To include CENTREID (labelled as INVID), subject no., randomisation no., period, randomised treatment, actual treatment and deviation. Also include PTYN and PTSUBJID from DMDATA.PRVTRIAL. | SAC |
| 2. | Screened<br>(Part A) | EX4 | Listing of Exposure Data (Single Dose) | Dose: extract from actual treatment (if dosing not completed, set to max. possible dose that could have been taken & include footnote). Exclude 'Cumulative Dose' and replace with 'No. Of Inhalations'. | SAC |
| Dispos | ition | | | | |
| 3. | Screened<br>(Part A) | CP_ES10x | Listing of Reasons for Withdrawal (Single Dose) | | SAC |
| 4. | Screened<br>(Part A) | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Single Dose) | | SAC |
| 5. | Screened<br>(Part A) | DV2 | Listing of Protocol Deviations (Single Dose) | | SAC |
| 6. | Screened<br>(Part A) | BL2 | Listing of Subjects For Whom the Treatment Blind was Broken (Single Dose) | | SAC |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphy | | | | |
| 7. | Screened<br>(Part A) | DM4 | Listing of Demographic Characteristics (Single Dose) | | SAC |
| 8. | Screened<br>(Part A) | DM10 | Listing of Race (Single Dose) | | SAC |
| Conco | mitant Medicati | ons and Adverse | Events | | |
| 9. | Screened<br>(Part A) | CP_CM4 | Listing of Concomitant Medications by Generic Term (Single Dose) | | SAC |
| 10. | Screened<br>(Part A) | CP_AE9 | Listing of All Adverse Events (Single Dose) | | SAC |
| 11. | Screened<br>(Part A) | CP_AE9a | Listing of Serious Adverse Events (Single Dose) | | SAC |
| 12. | Screened<br>(Part A) | AE7 | Listing of Subject Numbers for Individual Adverse Events (Single Dose) | | SAC |
| 13. | Screened<br>(Part A) | CP_AE9 | Listing of Adverse Events Leading to Withdrawal from Study (Single Dose) | | SAC |
| Safety | Assessments | | | | |
| 14. | Screened<br>(Part A) | CP_LB6 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance (Single Dose) | | SAC |
| 15. | Screened<br>(Part A) | CP_LB6 | Listing of All Clinical Chemistry Laboratory Data for Subjects with any Abnormality of Potential Clinical Importance (Single Dose) | | SAC |
| 16. | Screened<br>(Part A) | CP_LB6 | Listing of Haematology Abnormalities of Potential Clinical Importance (Single Dose) | | SAC |
| 17. | Screened<br>(Part A) | CP_LB6 | Listing of All Haematology Laboratory Data for Subjects with any Abnormality of Potential Clinical Importance (Single Dose) | | SAC |
| 18. | Screened<br>(Part A) | CP_VS5 | Listing of Vital Signs of Potential Clinical Importance (Single Dose) | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 19. | Screened<br>(Part A) | CP_VS5 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance (Single Dose) | | SAC |
| 20. | Screened<br>(Part A) | CP_EG4 | Listing of All 12-Lead ECG Values of Potential Clinical Importance (Single Dose) | | SAC |
| 21. | Screened<br>(Part A) | CP_EG4 | Listing of All 12-Lead ECG Values for Subjects with any Value of Potential Clinical Importance (Single Dose) | | SAC |
| 22. | Screened<br>(Part A) | CP_EG6 | Listing of Abnormal 12-Lead ECG Findings (Single Dose) | Clin sig change from baseline should not be populated for screening and pre-dose timepoints | SAC |
| 23. | Screened<br>(Part A) | UR2b | Listing of All Urinalysis Data (Single Dose) | | SAC |

# 10.11.12. ICH Listings: Part B (Repeat Dose)

| ICH : L | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Treatm | Treatment Information | | | | |
| 24. | Screened<br>(Part B) | CP_TA1 | Listing of Randomised and Actual Treatments (Repeat Dose) | To include CENTREID (labelled as INVID), subject no., randomisation no., randomised treatment, actual treatment and deviation | SAC |
| 25. | Screened<br>(Part B) | EX3 | Listing of Exposure Data (Repeat Dose) | Dose: extract from actual treatment (if dosing not completed, set to max. possible dose that could have been taken & include footnote). Include cumulative dose and insert extra column containing 'No. Of Inhalations'. | SAC |
| Dispos | ition | | | | |
| 26. | Screened<br>(Part B) | ES2 | Listing of Reasons for Withdrawal (Repeat Dose) | | SAC |
| 27. | Screened<br>(Part B) | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Repeat Dose) | | SAC |
| 28. | Screened<br>(Part B) | DV2 | Listing of Protocol Deviations (Repeat Dose) | | SAC |
| 29. | Screened<br>(Part B) | BL1 | Listing of Subjects For Whom the Treatment Blind was Broken (Repeat Dose) | | SAC |
| Demog | raphy | | | | |
| 30. | Screened<br>(Part B) | DM2 | Listing of Demographic Characteristics (Repeat Dose) | | SAC |
| 31. | Screened<br>(Part B) | DM9 | Listing of Race (Repeat Dose) | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Concor | mitant Medicati | ons and Adverse | Events | | • |
| 32. | Screened<br>(Part B) | CP_CM3 | Listing of Concomitant Medications by Generic Term (Repeat Dose) | | SAC |
| 33. | Screened<br>(Part B) | CP_AE8 (Part<br>B) | Listing of All Adverse Events (Repeat Dose) | | SAC |
| 34. | Screened<br>(Part B) | CP_AE8a (Part<br>B) | Listing of Serious Adverse Events (Repeat Dose) | | SAC |
| 35. | Screened<br>(Part B) | AE7 (Part B) | Listing of Subject Numbers for Individual Adverse Events (Repeat Dose) | | SAC |
| 36. | Screened<br>(Part B) | CP_AE8 (Part<br>B) | Listing of Adverse Events Leading to Withdrawal from Study (Repeat Dose) | | SAC |
| Safety | Assessments | | | | • |
| 37. | Screened<br>(Part B) | CP_LB5 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance (Repeat Dose) | | SAC |
| 38. | Screened<br>(Part B) | CP_LB5 | Listing of All Clinical Chemistry Laboratory Data for Subjects with any Abnormality of Potential Clinical Importance (Repeat Dose) | | SAC |
| 39. | Screened<br>(Part B) | CP_LB5 | Listing of Haematology Abnormalities of Potential Clinical Importance (Repeat Dose) | | SAC |
| 40. | Screened<br>(Part B) | CP_LB5 | Listing of All Haematology Laboratory Data for Subjects with any Abnormality of Potential Clinical Importance (Repeat Dose) | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 41. | Screened<br>(Part B) | CP_VS4 | Listing of Vital Signs of Potential Clinical Importance (Repeat Dose) | | SAC |
| 42. | Screened<br>(Part B) | CP_VS4 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance (Repeat Dose) | | SAC |
| 43. | Screened<br>(Part B) | CP_EG3 | Listing of All 12-Lead ECG Values of Potential Clinical Importance (Repeat Dose) | | SAC |
| 44. | Screened<br>(Part B) | CP_EG3 | Listing of All 12-Lead ECG Values for Subjects with any Value of Potential Clinical Importance (Repeat Dose) | | SAC |
| 45. | Screened<br>(Part B) | CP_EG5 | Listing of Abnormal 12-Lead ECG findings (Repeat Dose) | | SAC |
| 46. | Screened<br>(Part B) | UR2a | Listing of All Urinalysis Data (Repeat Dose) | | SAC |

# 10.11.13. Non-ICH Listings: Part A (Single Dose Escalation)

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | Data | | | | |
| 47. | Screened<br>(Part A) | AE2 | Relationship between System Organ Class and Verbatim Text (Single Dose) | | SAC |
| 48. | Screened<br>(Part A) | Other Listing 3<br>in<br>/arenv/arprod/g<br>sk2269557/pii1<br>15117/part_a/dr<br>ivers/saf_l3_cp<br>_hm7.sas | Listing of 24 Hour Holter Findings at Screening (Single Dose) | | SAC |
| 49. | Screened<br>(Part A) | Other Listing 2<br>in<br>/arenv/arprod/g<br>sk2269557/pii1<br>15117/part_a/dr<br>ivers/saf_I2_list.<br>sas | Listing of Cardiac Telemetry ECG Findings (Single Dose) | | SAC |
| Pharma | codynamic Da | ta | | | |
| 50. | Screened<br>(Part A) | PFT11 | Listing of %Predicted FEV1 Data at Screening (Single Dose) | To include 'Pred. Normal' and<br>'%Pred Normal' columns. Exclude<br>'Pre/Post Broncho' and '%Rev'<br>columns | SAC |
| 51. | Screened<br>(Part A) | PFT9 | Listing of FEV1 Data (Single Dose) | Include triplicate and maximum values. | SAC |

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 52. | Screened<br>(Part A) | Listing 63 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/part_c/dr<br>ivers/l_sputprep<br>_partc.sas | Listing of Sputum Sample Preparation and Haemacytometry/Cytospin Preparation Data (Single Dose) | Include sputum weight and time to first induction at each timepoint | SAC |
| 53. | Screened<br>(Part A) | Listing 64 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/part_c/dr<br>ivers/l_pip_part<br>c.sas | Listing of Phospholipid Data in Sputum (Single Dose) | | SAC |
| Pharma | cokinetic Data | l | | | |
| 54. | PK (Part A) | PKCL1x | Listing of Plasma GSK2292767 Pharmacokinetic Concentration-<br>Time Data (Single Dose) | | SAC |
| 55. | PK (Part A) | PKUL2x | Listing of Urine GSK2292767 Excretion Data(Single Dose) | Highest dose only so will only be 1 period of data | SAC |
| 56. | PK (Part A) | PKPL1x | Listing of Derived Plasma GSK2292767 Pharmacokinetic Data (Single Dose) | List all Part A PK parameters | SAC |

# 10.11.14. Non-ICH Listings: Part B (Repeat Dose)

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | Data | | | | |
| 57. | Screened<br>(Part B) | AE2 | Relationship between System Organ Class and Verbatim Text (Repeat Dose) | | SAC |
| 58. | Screened<br>(Part B) | Other Listing 3<br>in<br>/arenv/arprod/g<br>sk2269557/pii1<br>15117/part_a/dr<br>ivers/saf_l3_cp<br>_hm7.sas | Listing of 24 Hour Holter Findings at Screening (Repeat Dose) | | SAC |
| 59. | Screened<br>(Part B) | Similar to Other<br>Listing 2 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>15117/part_a/dr<br>ivers/saf_I2_list.<br>sas | Listing of Cardiac Telemetry ECG Findings (Repeat Dose) | According to the protocol, cardiac telemetry might also be done in Part B depending on emerging data. | SAC |
| Pharma | acodynamic Da | ta | | | |
| 60. | Screened<br>(Part B) | PFT11 | Listing of %Predicted FEV1 Data at Screening (Repeat Dose) | To include 'Pred. Normal' and<br>'%Pred Normal' columns. Exclude<br>'Pre/Post Broncho' and '%Rev'<br>columns | SAC |
| 61. | Screened<br>(Part B) | PFT8 | Listing of FEV1 Data (Repeat Dose) | Include triplicate and maximum values. | SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 62. | Screened<br>(Part B) | Listing 100 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/part_b/dr<br>ivers/l_sputprep<br>_partb.sas | Listing of Sputum Sample Preparation and Haemacytometry/Cytospin Preparation Data (Repeat Dose) | Include sputum weight and time to first induction at each timepoint | SAC |
| 63. | Screened<br>(Part B) | Listing 102 in /arenv/arprod/g sk2269557/pii1 16617/part_b/dr ivers/l_pip_part b.sas | Listing of Phospholipid Data in Sputum (Repeat Dose) | | SAC |
| Pharma | acokinetic Data | l | | | |
| 64. | PK (Part B) | PKCL1p | Listing of Plasma GSK2292767 Pharmacokinetic Concentration-<br>Time Data (Repeat Dose) | | SAC |
| 65. | PK (Part B) | PKPL1p | Listing of Derived Plasma GSK2292767 Pharmacokinetic Parameters (Repeat Dose) | | SAC |
| 66. | PK (Part B) | Listing 94 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/parts_cb<br>/drivers/l_pkacc<br>um_partcb.sas | Listing of Peak and Trough Accumulation and GSK2292767 Peak:Trough Ratios (Repeat Dose) | | SAC |

| Non-IC | Non-ICH: Listings | | | |
|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title Programming Notes | Deliverable<br>[Priority] |
| 67. | PK (Part B) | Listing 98 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/part_b/dr<br>ivers/nich_l98_<br>part_b.sas | Listing of Plasma and BAL Fluid Urea Data (Repeat Dose) Include Dilution Factor | SAC |
| 68. | PK (Part B) | Listing 99 in<br>/arenv/arprod/g<br>sk2269557/pii1<br>16617/part_b/dr<br>ivers/nich_l99_<br>partb.sas | Listing of BAL Fluid and Derived Lung ELF GSK2292767 Pharmacokinetic Concentration Data (Repeat Dose) Include Dilution Factor and variables in Example output. Include footnote for BAL Fluid Councentrations instead of raw concentrations. | - Δ(: |